CLINICAL TRIAL: NCT07035132
Title: Effects of the Specific Supplementation (100% Seric Hydrolized Lactoprotein and MCT) in Malnourished Oncologic Patients Undergoing Radiotherapy
Brief Title: Impact of Specific Oligomeric Supplementation in Oncologic Patients Undergoing Radiotherapy With Malnutrition or at Risk.
Acronym: NORMA
Status: Enrolling by invitation | Type: Observational
Sponsor: Outcomes'10 (Network)
Collaborators: Nestlé Health Science Spain (Industry)
Responsible Party: Sponsor
Other Study IDs: NES-2023-154-PRO-PEP
Record Dates: First submitted 2025-05-15; First posted 2025-06-24 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Malnutrition in Elderly; Oncological Patients; Digestive Disorders
Keywords: nutritional supplementation; radiotherapy; malabsortion; oligomeric formula
MeSH Terms: conditions — Digestive System Diseases | interventions — Dietary Supplements

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Oral supplementation with nutritional oligomeric formula — Patients will be supplemented with the specific oligomeric formula (1 or 2 bottles/day, as per investigator's decision) during, at least, the 12 weeks of the study follow-up.

SUMMARY:
An observational, prospective, multicenter study to be conducted in 5 hospitals in Spain. Patients with cancer undergoing radiotherapy are malnourished or at risk of malnutrition. Due to the characteristics of their pathology or gastrointestinal disorders, the use of oligomeric nutritional formulas formulated with 100% hydrolyzed whey lactoprotein and a high MCT content is recommended as part of routine clinical practice. Patients will be followed for 12 weeks, with three visits: a baseline visit upon inclusion in the study, after 6 weeks and a final visit 12 weeks after the nutritional treatment starts.

DETAILED DESCRIPTION:
The prevalence of malnutrition is high in cancer patients: about 80% of patients will suffer from malnutrition at some point, and it is the cause of 10-20% of deaths in this type of patient.

To address malnutrition in these patients, international clinical guidelines recommend periodically reviewing their nutritional status and supplementing with oral nutrition formulas (ONS) when they are unable to meet their nutritional needs from their usual diet.

The ONSs have a nutrient composition designed to meet the specific needs of the patient, but there are pathologies, types of tumours and treatments, such as radiotherapy, chemotherapy, immunotherapy and others that can alter the digestion process, making it difficult for the gastrointestinal tract to utilise nutrients. Patients with these pathologies often cannot tolerate polymeric SNO formulations and require oligomeric peptide-based diet (PBD) formulations.

PBDs contain hydrolysed proteins in the form of peptides and medium-chain triglycerides (MCTs), which are more easily assimilated, helping patients to reduce weight loss and improve overall nutritional status. In addition, they contain hydrolysed serum lactoprotein with high biological quality that stimulates the formation of muscle tissue, minimising cachexia.

Radio/chemotherapy/immunotherapy treatment has negative effects on the nutritional and functional status of cancer patients, which also makes them more susceptible to the toxicities of cancer treatments and clinical complications. It has been shown that these patients tolerate PBD formulas well and even reduce their baseline intestinal symptoms, which facilitates compliance with nutritional treatment. However, adherence to these treatments remains a challenge as it is not always optimal, resulting in the non-achievement of the potential benefits.

The main objective of the study is to evaluate the effects of a hypercaloric SNO, with 100% hydrolysed serum lactoprotein and high MCT intake, in cancer patients undergoing radiotherapy, malnourished or at risk of malnutrition, in terms of improving the patient's nutritional status after 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients of legal age (≥18 years).
* Oncology patients (with head and neck, lung or rectal cancer) undergoing or about to start radiotherapy treatment. Patients with oesophageal cancer will also be included, as long as the patient is not undergoing PEG.
* Patients who are malnourished or at risk of malnutrition according to GLIM criteria.
* Patients requiring supplementation with an oligomeric formula with 100% hydrolysed serum lactoprotein and high MCT intake due to gastrointestinal disturbances (either maldigestion or maldigestion, malabsorption or dysmotility) intolerance to polymeric formulations or any other reason as considered by the physician.
* Patients who, at the discretion of the investigator, have the ability to answer the questionnaires and follow the procedures detailed in the protocol.
* Patients who give written informed consent to participate.

Exclusion Criteria:

* Patients with galactosemia, allergies and/or intolerances to lactose or any of the compounds of the formula.
* Patients receiving nutritional support other than that of the study characteristics or who have received it during the last month. It will be accepted in patients who, being on a polymeric SNO, are advised to change to the oligomeric formula under study, due to gastrointestinal alterations, intolerances or any other reason considered by the doctor.
* Patients who have undergone surgery in the last three months.
* Patients who have received Enteral Nutrition in the last 3 months for SNG/SNJ/PEG.
* Pregnant or lactating women.
* Patients with advanced renal or hepatic disease (with creatinine clearance less than 45 ml/min or CP=C).
* Patients with advanced neoplastic disease with life expectancy <3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oncological patients undergoing radiotherapy, who present malnutrition or risk of malnutrition and due to the characteristics of the pathology or gastrointestinal alterations, the use of oligolimeric nutritional formulas formulated with 100% hydrolyzed serum lactoprotein and high MCT content is recommended within the usual clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who improve the degree of malnutrition. | From enrollment to the end of treatment at 12 weeks
  According to body weight, after 12 weeks of treatment with SNO with 100% hydrolyzed serum lactoprotein and high MCT intake.

SECONDARY OUTCOMES:
Percentage of patients with improvement in the degree of malnutrition | From enrollment to the end of treatment at 12 weeks
  According to GLIM criteria after 12 weeks of treatment with SNO with 100% hydrolyzed serum lactoprotein and high MCT intake.
Percentage change in BMI | From enrollment to the end of treatment at 12 weeks
  Weight and height will be combined to report BMI in kg/m².
Arm circumference | From enrollment to the end of treatment at 12 weeks
  Is measured in CM
Calf circumference | From enrollment to the end of treatment at 12 weeks
  Is measured in CM
Maximum prehensile strength value | From enrollment to the end of treatment at 12 weeks
  Using a dynamometer, an instrument that measures force in kilograms.
Sit-to-stand test | From enrollment to the end of treatment at 12 weeks
  Is measured primarily by counting the number of repetitions a person can perform while standing up and sitting in a chair in a specified period of time, such as 30 seconds.
Impedancemetry values | From enrollment to the end of treatment at 12 weeks
  Probe.
Percentage of patients presenting complications associated with nutritional status during treatment. | From enrollment to the end of treatment at 12 weeks
  Changes in oncological treatment, hospital admissions or visits to the emergency room are considered complications.
Percentage of patients presenting changes in gastrointestinal tolerance after 6 and after 12 weeks of treatment with SNO with 100% hydrolyzed serum | After 6 and after 12 weeks of treatment
  After 6 and after 12 weeks of treatment with SNO with 100% hydrolyzed serum lactoprotein and high MCT intake.
Distribution of the patients according to their compliance with the treatment | At 6 and 12 weeks of treatment.
  With SNO with 100% hydrolyzed serum lactoprotein and high MCT intake.
Distribution of the patients according to their adherence to the treatment | At 6 and 12 weeks of treatment.
  (low: 0-2 points, medium: 3-4 points or high: 5-6 points)
Percentage of patients who maintain or improve their quality of life after 12 weeks of treatment. | After 12 weeks of treatment.
  Improve their quality of life.
Percentage of patients satisfied with the product | After 12 weeks of treatment with SNO
  With SNO with 100% hydrolyzed serum lactoprotein and high MCT content.
Average health care expenditure per patient, according to degree of malnutrition, during the study. | From enrollment to the end of treatment at 12 weeks
  Health expenditure per patient

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Hospital Universitario San Juan de Alicante, Alicante
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - HU Clinica Asturias, Oviedo
  - Hospital Universitario Son Espases, Palma de Mallorca

IPD SHARING:
Plan to Share IPD: No